CLINICAL TRIAL: NCT05609695
Title: Immune Checkpoint Inhibitor Monotherapy or Combined With Molecular Targeted Drugs / Locoregional Therapy in the Treatment of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Chief physician, Sun Yat-sen University
Other Study IDs: B2022-341-01
Record Dates: First submitted 2022-11-03; First posted 2022-11-08 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Immune Checkpoint Inhibitor Monotherapy or Combined With Molecular Targeting Drugs / Locoregional Therapy for Hepatocellular Carcinoma
Keywords: Immune checkpoint inhibitor; locoregional therapy; combination therapy; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Immunotherapy group: Treatment based on immunotherapy.
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — After signing the written informed consent form, patients begin to receive single or combined therapy with immune checkpoint inhibitor. The use of immune checkpoint inhibitors takes 3 weeks as a cycle, and the treatment dose for each cycle is carried out in accordance with the latest international authoritative guidelines.

SUMMARY:
Non-intervention observation to evaluate the safety and efficacy of immune checkpoint inhibitors alone or combined with molecular targeted drugs / local interventional therapy in patients with advanced liver cancer, and to provide the best choice for the treatment of patients with advanced liver cancer in different stages.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures.
2. Cytohistological confirmation is required for diagnosis of HCC.
3. Patients with advanced (unresectable and/or metastatic, stage C based on Barcelona-Clinic Liver Cancer [BCLC] staging classification) hepatocellular carcinoma which would not be suitable for treatment with loco-regional therapies or have progressed following locoregional therapy such as surgical resection, percutaneous hepatic arterial embolization, radiofrequency ablation, and percutaneous interventional therapy.
4. At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.
5. Current cirrhotic status of Child-Pugh class A-B, with no encephalopathy. Ascites controlled by diuretics is permitted in this study.
6. Availability of a representative tumor tissue specimen (archival tumor tissue is allowed) at pre-screening.
7. astern Cooperative Oncology Group Scale for Assessment of Patient Performance Status ≤ 2.
8. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial.
9. Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to procedure:

   Hemoglobin > 100g/L Absolute neutrophil count >3.0 ×109/L Neutrophil count > 1.5 ×109/L Platelet count ≥ 50.0 ×109/L Total bilirubin < 51 μmol/L Alanine transaminase (ALT) and aminotransferase (AST) < 5 x upper limit of normal Albumin > 28 g/L Prothrombin time (PT)-international normalized ratio (INR) < 2.3, or PT < 6 seconds above control Serum creatinine < 110 μmol/L
10. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Received any prior systemic chemotherapy or molecular-targeted therapy for HCC such as sorafenib, lenvatinib.
2. Previous local therapy completed less than 4 weeks prior to the dosing and, if present any related acute toxicity > grade 1.
3. Any contraindications for Immune checkpoint inhibitor procedure
4. Renal failure / insufficiency requiring hemo-or peritoneal dialysis.
5. Known severe atheromatosis.
6. Known uncontrolled blood hypertension (> 160/100 mm/Hg).
7. Patients with any other malignancies within the last 3 years before study start.
8. History of HCC tumor rupture.
9. Patients with severe encephalopathy. Patients with known active bleeding (e.g. from GI ulcers, esophageal varices) within 2 months prior to baseline/screening visit or with history or evidence of inherited bleeding diathesis or coagulopathy.
10. History of cardiac disease.
11. Any other condition that would, in the Investigator's judgment, contraindicate patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable or unwilling to swallow medication, social/ psychological issues, etc.
12. Patients who have received any other investigational agents within a period of time that is less than the cycle length used for that treatment or equal to 4 weeks (whichever is shorter) prior to starting study drug and recovered from any side effects to grade 1 or less.
13. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients aged from 18 to 75 years old were diagnosed as hepatocellular carcinoma by pathological diagnosis and were in stage C of BCLC.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3-years Followed up
  Absence of death of any cause

SECONDARY OUTCOMES:
Tumor Response | 3-years Followed up
  Tumor response to immune checkpoint inhibitor according to RECIST 1.1
Progress Free Survival | 3-years Followed up
  Absence of disease progression other than death

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, M.D. & Ph.D., Principal Investigator — Department of Minimally Invasive and Interventional Radiology, Liver Cancer
Locations (1):
- Department of Minimally Invasive and Interventional Radiology, Liver Cancer Study and Service Group, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lyu N, Wang X, Li JB, Lai JF, Chen QF, Li SL, Deng HJ, He M, Mu LW, Zhao M. Arterial Chemotherapy of Oxaliplatin Plus Fluorouracil Versus Sorafenib in Advanced Hepatocellular Carcinoma: A Biomolecular Exploratory, Randomized, Phase III Trial (FOHAIC-1). J Clin Oncol. 2022 Feb 10;40(5):468-480. doi: 10.1200/JCO.21.01963. Epub 2021 Dec 14. PMID 34905388
- [Result] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013